CLINICAL TRIAL: NCT05751642
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Study of Subcutaneously and Intravenously Administered ALXN1920 in Healthy Adult Participants
Brief Title: Safety and Tolerability, Pharmacokinetic, and Pharmacodynamic Study of ALXN1920 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: ALXN1920-HV-101
Record Dates: First submitted 2023-02-21; First posted 2023-03-02 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Healthy Participants
Keywords: First-in-human; Single ascending dose; Sentinel dosing; ALXN1920; Safety; Pharmacokinetics; Pharmacodynamics; Japanese Descent

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Cohort 1 (Experimental): Participants will receive a single dose of ALXN1920.
  Interventions: Biological: ALXN1920
- Cohort 2 (Experimental): Participants will receive a single dose of ALXN1920.
  Interventions: Biological: ALXN1920
- Cohort 3 (Experimental): Participants will receive a single dose of ALXN1920.
  Interventions: Biological: ALXN1920
- Cohort 4 (Experimental): Participants will receive a single dose of ALXN1920.
  Interventions: Biological: ALXN1920
- Cohort 5 (Experimental): Participants will receive a single dose of ALXN1920.
  Interventions: Biological: ALXN1920
- Cohort 6: Japanese Cohort (Experimental): Japanese participants will receive a single dose of ALXN1920.
  Interventions: Biological: ALXN1920
- Pooled Placebo (Placebo Comparator): Participants will receive Placebo.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: ALXN1920 — Participants will receive a single dose of ALXN1920 by Subcutaneous (SC) injection.
  Arms: Cohort 1; Cohort 2
Biological: Placebo — Participants will receive a single dose of Placebo by SC injection, SC infusion or IV infusion.
  Arms: Pooled Placebo
Biological: ALXN1920 — Participants will receive a single dose of ALXN1920 by SC infusion.
  Arms: Cohort 3; Cohort 4; Cohort 6: Japanese Cohort
Biological: ALXN1920 — Participants will receive a single dose of ALXN1920 by Intravenous (IV) infusion.
  Arms: Cohort 5

SUMMARY:
This study will assess the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and immunogenicity of single ascending doses (SADs) of ALXN1920 subcutaneous (SC) and of a single dose of ALXN1920 intravenous (IV) in healthy adult participants.

DETAILED DESCRIPTION:
This is a first-in-human study in healthy adult participants.

Eligible participants will be randomly assigned in a 3:1 (ALXN1920:Placebo) ratio in each of the treatment cohorts. The first 2 participants randomized to each cohort will be dosed as a sentinel pair, with 1 participant on active treatment and 1 participant on placebo. At the discretion of the Investigator, up to 3 more participants will be added at least 48 hours after the dosing of the sentinel pair, followed by dosing of the remaining participants in the cohort no earlier than 72 hours after sentinel pair dosing.

The study will comprise:

A Screening Period of up to 28 days; A Dosing Period (single dose through to Follow-up Visit) of approximately 28 days; A Final Follow-up period and end of study Visit is planned on Day 29.

Each participant will be involved in the study for approximately 56 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants
* Body mass index within 18.0 to 32.0 kg/m^2 (inclusive), with a minimum body weight of 50.0 kg.
* Female participants of childbearing potential and male participants must follow protocol-specified contraception guidance.
* For Cohort 6, participants of Japanese descent, defined as having both parents and 4 grandparents who are ethnically Japanese.

Exclusion Criteria:

* Significant history or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, or neurological disorders.
* History of significant allergic reaction.
* History of any Neisseria infection
* Active systemic bacterial, viral, or fungal infection.
* Participants who at Day -1 are either testing positive for coronavirus disease 2019 (COVID-19), or have not had at least 4 weeks elapse of recovery time (a negative test), or are experiencing long-term COVID-19-related sequelae.
* Any major surgery within 8 weeks of Screening.
* Known or suspected history of drug or alcohol abuse.
* Current tobacco users or smokers.
* Positive Human immunodeficiency virus (HIV) infection, hepatitis B or hepatitis C viral infection.
* Female participant who are pregnant, breastfeeding, or intending to conceive during the course of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2023-04-19 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2023-12-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse events (AEs) | Up to End of study visit (Day 29)
  To assess the safety and tolerability of single ascending doses of ALXN1920.

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) | Day 1 (Pre-dose, 0.5, 1, 2, 6 and 12 hours post-dose), post-dose on Day 2, 3, 4, 5, 6, 8, 15, 22, and 29
  To assess the Cmax of ALXN1920 following single ascending doses of ALXN1920.
Time to maximum observed concentration (tmax) | Day 1 (Pre-dose, 0.5, 1, 2, 6 and 12 hours post-dose), post-dose on Day 2, 3, 4, 5, 6, 8, 15, 22, and 29
  To assess the tmax of ALXN1920 following single ascending doses of ALXN1920.
Area under the concentration-time curve from time 0 (dosing) to the last quantifiable concentration (AUC0-t) | Day 1 (Pre-dose, 0.5, 1, 2, 6 and 12 hours post-dose), post-dose on Day 2, 3, 4, 5, 6, 8, 15, 22, and 29
  To assess the AUC0-t of ALXN1920 following single ascending doses of ALXN1920.
Area under the concentration-time curve from time 0 (dosing) to time infinity (AUCinf) | Day 1 (Pre-dose, 0.5, 1, 2, 6 and 12 hours post-dose), post-dose on Day 2, 3, 4, 5, 6, 8, 15, 22, and 29
  To assess the AUCinf of ALXN1920 following single ascending doses of ALXN1920.
Terminal elimination half-life (t½) | Day 1 (Pre-dose, 0.5, 1, 2, 6 and 12 hours post-dose), post-dose on Day 2, 3, 4, 5, 6, 8, 15, 22, and 29
  To assess the t½ of ALXN1920 following single ascending doses of ALXN1920.
Terminal-phase elimination rate constant (λz) | Day 1 (Pre-dose, 0.5, 1, 2, 6 and 12 hours post-dose), post-dose on Day 2, 3, 4, 5, 6, 8, 15, 22, and 29
  To assess the λz of ALXN1920 following single ascending doses of ALXN1920.
Total body clearance (CL) | Day 1 (Pre-dose, 0.5, 1, 2, 6 and 12 hours post-dose), post-dose on Day 2, 3, 4, 5, 6, 8, 15, 22, and 29
  To assess the CL of ALXN1920 following single ascending doses of ALXN1920.
Apparent clearance (CL/F) | Day 1 (Pre-dose, 0.5, 1, 2, 6 and 12 hours post-dose), post-dose on Day 2, 3, 4, 5, 6, 8, 15, 22, and 29
  To assess the CL/F of ALXN1920 following single ascending doses of ALXN1920.
Volume of distribution (Vd) | Day 1 (Pre-dose, 0.5, 1, 2, 6 and 12 hours post-dose), post-dose on Day 2, 3, 4, 5, 6, 8, 15, 22, and 29
  To assess the Vd of ALXN1920 following single ascending doses of ALXN1920.
Apparent volume of distribution (Vd/F) | Day 1 (Pre-dose, 0.5, 1, 2, 6 and 12 hours post-dose), post-dose on Day 2, 3, 4, 5, 6, 8, 15, 22, and 29
  To assess the Vd/F of ALXN1920 following single ascending doses of ALXN1920.
Renal clearance (CLR) | Day 1 through Day 5 (Pre-dose and up to 96 hours post-dose)
  To assess the CLR of ALXN1920 following single ascending doses of ALXN1920.
Amount of unchanged drug excreted in urine (Ae) | Day 1 through Day 5 (Pre-dose and up to 96 hours post-dose)
  To assess the Ae of ALXN1920 following single ascending doses of ALXN1920.
Fraction of dose excreted in urine (fe) | Day 1 through Day 5 (Pre-dose and up to 96 hours post-dose)
  To assess the fe of ALXN1920 following single ascending doses of ALXN1920.
Change in complement alternative pathway (CAP) activity | Day 1 (Pre-dose, 0.5, 1 and 2 hours post-dose), post-dose on Day 2, 3, 4, 5, 8, 15, 22, and 29
  To explore the Pharmacodynamic (PD) effects of single ascending doses of ALXN1920. CAP activity will be assessed using the CAP hemolytic assay.
Change in factor H | Day 1 (Pre-dose, 0.5, 1 and 2 hours post-dose), post-dose on Day 2, 3, 4, 5, 8, 15, 22, and 29
  To explore the PD effects of single ascending doses of ALXN1920. Change in factor H will be assessed using the factor H assay.
Number of Participants With Positive Antidrug Antibodies (ADAs) to ALXN1920 | Day 1 pre-dose and Day 29 post-dose
  To assess the immunogenicity to ALXN1920.
Geometric Mean Ratio (GMR) of Area Under the Curve (AUC) Values of Subcutaneous (SC) Versus Intravenous (IV) Serum Concentration of ALXN1920 | Day 29 post-dose
  To assess the absolute bioavailability of ALXN1920 SC.

CONTACTS AND LOCATIONS:
Locations (2):
- New Zealand (2):
  - Clinical Trial Site, Grafton, Auckland
  - Research Site, Christchurch

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home